CLINICAL TRIAL: NCT00632723
Title: A Phase II Trial to Assess the Efficacy of IRESSA™ (Gefitinib) 500 mg/Day in Patients With Breast Cancer Who Have Failed Tamoxifen or Have an Oestrogen Receptor Negative Tumour and Would be Considered for Systemic Therapy
Brief Title: IRESSA™ (Gefitinib) in Breast Cancer Patients
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Pauline Pert, Clinical Leader, AZ UK MC, AstraZeneca
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1839IL/0057
Record Dates: First submitted 2008-01-17; First posted 2008-03-11 (Estimated); Last update posted 2009-04-22 (Estimated); Status verified 2009-04

CONDITIONS: Breast Cancer
Keywords: oestrogen receptor; ER negative tumours; epidermal growth factor receptor (EGFR)
MeSH Terms: conditions — Breast Neoplasms | interventions — Gefitinib

INTERVENTIONS:
Drug: gefitinib (IRESSA™, ZD1839) — 250 mg tablet; daily dose 500 mg daily
  Other Names: IRESSA™; ZD1839

SUMMARY:
This is a phase II trial to assess whether IRESSA™ (gefitinib) has anti-tumour efficacy in patients with breast cancer. The trial proposes to enter 27 patients who have acquired resistance to tamoxifen and 27 patients with ER negative tumours. However for each of these two types of patients recruitment will stop after 14 patients have been entered in order to confirm that IRESSA™ (gefitinib)has anti-tumour efficacy. If no patient out of 14 in a group has shown clinical benefit (ie an objective response (CR or PR) or stable disease (SD) for at least 24 weeks) then a clinical benefit rate of >20% can be ruled out with >95% certainty. If one or more of the objective response or stable disease (> 24 weeks) has been seen in the first 14 patients recruited in a group then recruitment to that group will recommence to a total of 27 patients. If 14 patients are entered into an arm but not all 14 patients are available for final analysis and the toxicity/safety and tolerability profile of the therapy is acceptable and documented and a clinical benefit is seen in the patients, enrolment of additional patients beyond the initial 14 may be made based on overall clinical assessment.

ELIGIBILITY:
Inclusion Criteria:

* histological or cytological confirmation of breast cancer that is either

  * a primary tumour in a patient unfit for or who has declined surgery
  * advanced (locally or metastatic) disease
* acquired resistance to tamoxifen or ER negative tumour
* at least one measurable or assessable lesion
* WHO performance status 0 - 2
* life expectancy of 12 weeks or more

Exclusion Criteria:

* more than one previous chemotherapy regimens for advanced disease
* prior anthracycline chemotherapy (> 250 mg/m2 adriamycin)
* radiotherapy completed within 14 days prior to Day 1 of treatment
* incomplete healing from prior oncologic or other major surgery
* signs of neurological symptoms consistent with spinal cord compression
* any evidence of clinically active interstitial lung disease (patients with chronic stable

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 54 (Actual)
Dates: Start 2001-04; Study Completion 2005-10 (Actual)

PRIMARY OUTCOMES:
Objective tumour response (complete + partial response) based on Union International Contre le Cancer (UICC) Criteria | Assessed after 24 weeks
Clinical benefit (CR + PR + SD > 24 wks) | After 24 weeks of treatment
Frequency and severity of adverse events (AEs) | Assessed at each visit

SECONDARY OUTCOMES:
Progression-free survival | Time to death
Duration of response | Time to progression

CONTACTS AND LOCATIONS:
Overall Officials: R Robertson, MD, Principal Investigator — City Hospital, Nottingham , UK